CLINICAL TRIAL: NCT02742636
Title: When is the Best Moment to Remove the Urinary Catheter After Laparoscopic Hysterectomy: MUCH Study.
Brief Title: When is the Best Moment to Remove the Urinary Catheter After Laparoscopic Hysterectomy?
Acronym: MUCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Bronovo Hospital (Other); Haga Hospital (Other); Alrijne Hospital (Other); Reinier de Graaf Groep (Other); Groene Hart Ziekenhuis (Other); Medical Center Haaglanden (Other)
Responsible Party: Principal Investigator, FWJansen, Prof. Dr, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P15.382
Record Dates: First submitted 2016-04-01; First posted 2016-04-19 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Urinary Tract Infection; Bladder Retention
MeSH Terms: conditions — Urinary Tract Infections; Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (treatment group) (Experimental): The patients in this group will have their catheter directly removed in the OR after LH.
  Interventions: Device: Foley catheter
- Group B (control group) (Active Comparator): The patients in the control group will have their catheter removed according to the regular protocol of the hospital (at least 6 hours in place).
  Interventions: Device: Foley catheter

INTERVENTIONS:
Device: Foley catheter — The aim of this study is to evaluate if direct removal of the urine catheter after an LH (total laparoscopic hysterectomy and laparoscopic supracervical hysterectomy) is associated with similar (or better) outcomes compared to delayed catheter removal after surgery.

SUMMARY:
Objective: The aim of this study is to evaluate if direct removal of the urine catheter after an laparoscopic hysterectomy (total laparoscopic hysterectomy and laparoscopic supracervical hysterectomy) is associated with similar (or better) outcomes compared to delayed catheter removal after surgery, which is the current treatment. In addition, we want to investigate patient's experience on this subject.

Study design: Randomized Controlled trial, non-inferiority study.

Study population: Women older than 18 years old, who are a laparoscopic hysterectomy for benign indication or low-grade malignancy.

Intervention:

* Group A (treatment group): the patients in this group will have their catheter directly removed in the OR after LH.
* Group B (control group): the patients in the control group will have their catheter removed according to the regular protocol of the hospital (at least 6 hours in place).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Scheduled for LH for benign indication or low-grade malignancy (with or without salpingo-oophorectomy)

Exclusion Criteria:

* Concomitant procedures such as prolapse surgery, severe endometrioses and/or bowel resection
* Preoperative known urinary voiding problems (incontinence)
* Preoperative known urinary tract infection
* Patients suffering from diseases potentially associated with inability to void (e.g. MS)
* A Gravid or postpartum hysterectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Urinary retention (inability to void) | 6 hours after removal of urinary catheter

SECONDARY OUTCOMES:
Rate of re-catheterisation | 6 hours without voiding
Urinary tract infection (by performing a urine dipstick test and based on clinical symptoms) | Dipstick: first urine after removal of catheter (group 1: direct after OR, group 2: at least 6 hours after OR), clinical symptoms through study period (up to 6 weeks postoperative)
Patient satisfaction (self-administrated questionnaire) | 6 hours postoperative; 24 hours and 6 weeks
Visual analogue scale score (VAS score) | 6 hours postoperative; 24 hours

CONTACTS AND LOCATIONS:
Locations (7):
- Netherlands (7):
  - Leiden University Medical Center, Leiden, North Holland
  - Reinier de Graaf Groep, Delft
  - Groene Hart Ziekenhuis, Gouda
  - Alrijne Hospital, Leiden
  - Bronovo Hospital, The Hague
  - Haga Hospital, The Hague
  - Medisch Centrum Haaglanden, The Hague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246